CLINICAL TRIAL: NCT06873191
Title: Post-Approval Safety Monitoring Program to Assess the Safety and Efficacy Profile of TUKYSA in Usual Practice
Brief Title: A Study to Learn More About Tukysa Once it is Out in the Korean Market
Status: Not yet recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C4251017
Record Dates: First submitted 2025-03-06; First posted 2025-03-12 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: HER2-positive Locally Advanced Unresectable; Metastatic Breast Cancer
Keywords: safety
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objectives of the re-examination system in Korea is to re-confirm the clinical usefulness of the product through collecting, reviewing, identifying and verifying the safety and efficacy information about the product in general practice in Korea.

This surveillance is conducted for preparing application material for re-examination under the Pharmaceutical Affairs Laws, the Regulations on Safety of Pharmaceuticals, etc. and the Re-examination Regulation for New Drugs and Others.

DETAILED DESCRIPTION:
The purpose of this study is to understand the safety of Tukysa (Tucatinib hemiethanolate) once it is out in the Korean market. Tukysa will be given to participants aged 18 or over in Republic of Korea.

Surveillance Design Patients with the approved indication who are treated with TUKYSA within the local label will be enrolled.

Adverse Events (AEs) will be collected in the usual practice during administration and for 28 days following cessation of TUKYSA, and ORR will be evaluated through radiographic imaging in the usual practice. The total follow-up period will not exceed 1 year.

Safety

Through the evaluation the safety profile of TUKYSA including important identified risks, Important potential risks, missing information, which are defined about TUKYSA in table2, will be examined. Drug safety is evaluated through the following items:

Efficacy Drug efficacy will be evaluated through the BOR. The ORR which is defined as the proportion of the subjects in the analysis population who have best response as CR or PR will be presented.

Surveillance for long-term use The follow-up period for each patient will vary according to tumor response, treatment of TUKYSA and others. Any patients who are treated with TUKYSA for more than or equal to 180 days including dose interruption will be evaluated for surveillance for long-term use.

ELIGIBILITY:
Inclusion criterias.

1. Patient who is treated with TUKYSA according to the current TUKYSA label for the approved indication.
2. Patient who is treated with TUKYSA for the first time.
3. Patient who is aged 18 or over.
4. Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study.

Exclusion criterias.

1. Patients to whom TUKYSA is contraindicated as per the local labeling Note: The summary for any patients who are violated in the inclusion/exclusion criteria (i.e. protocol violation case) will be separately done if collected and described in the separate section of the report.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population for this study includes subjects aged 18 years or older who will be monitored for any adverse events during treatment with TUKYSA® Tablets and for 28 days following the cessation of treatment in the Republic of Korea.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2027-01-01 (Estimated); Primary Completion 2029-05-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From Day 1 through Day 7 after administration. Administration and for 28 days following. The total follow-up period will not exceed 1 year.
  The BOR from the start of treatment until progressive disease (PD)/recurrence will be recorded in the electronic Case Report Form as CR, PR, stable disease (SD), PD or Not Evaluable (NE).
  The BOR will be defined the best overall response recorded from the start of treatment until PD/recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.